CLINICAL TRIAL: NCT04855994
Title: Comparison of the Results of Ultrasound-Guided Thoracic Paravertebral Block and Modified Pectoral Nerve Block for Postoperative Analgesia in Video-Assisted Thoracoscopic Surgery; A Prospective, Randomized Controlled Study
Brief Title: Comparison of Thoracic Paravertebral Block and Pectoral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Sertcakacilar, MD, Principal Investigator, MD, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-140
Record Dates: First submitted 2021-04-09; First posted 2021-04-22 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Thoracic Paravertebral Block; Video-assisted Thoracoscopic Surgery; Postoperative Analgesia
Keywords: Thoracic paravertebral block,; pectoralis block,; Video-assisted thoracoscopic surgery,; Postoperative analgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paravertebral group (Active Comparator): The investigators performed Paravertebral block to that patient group for postoperative analgesia
  Interventions: Procedure: paravertebral block
- pectoral group (Active Comparator): The investigators performed pectoral block to that patient group for postoperative analgesia
  Interventions: Procedure: pectoral block

INTERVENTIONS:
Procedure: paravertebral block — The investigators performed Paravertebral block to that patient group for postoperative analgesia
  Arms: paravertebral group
Procedure: pectoral block — The investigators performed pectoral block to that patient group for postoperative analgesia
  Arms: pectoral group

SUMMARY:
This study aims to compare the efficacy and safety of ultrasound-guidedPECS II block with TPVB for postoperative analgesia after VATS.

DETAILED DESCRIPTION:
52 patients (ASA I-III) between 18 and 65 years of age, who were to undergo VATS, were randomized and divided into two groups. (26 patients in each of the PECS and TPVB groups) Thoracic paravertebral block was administered from two consecutive levels for TPVB group and a modified pectoral nerve block was performed in the PECS group. Postoperative analgesia was provided by intravenous morphine infusion using a patient-controlled analgesia device. Postoperative 24-hour total morphine consumption and duration of analgesia were the primary outcome measure. Perioperative remifentanil use, visual analog scale values during at rest and coughing, time of the first analgesic request, and additional analgesic consumption were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-65
* Patients who will undergo VATS
* ASA I-II-III patients

Exclusion Criteria:

* Patients with ASA IV
* Clinically diagnosis of spinal or chest wall deformity or pathology
* Clinically known local anesthetic allergy
* Morbid obesity (body mass index>40 kg m2)
* Clinically diagnosis of opioid, alcohol and substance dependence
* Clinically diagnosis of psychiatric disease
* Coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Postoperative 24-hours total morphine consumption of patients | 24 hours postoperatively
  This will be measured only one time by pca device at the 24th hour after surgery.

SECONDARY OUTCOMES:
Visual Analog Scale values of patients | 24 hours postoperatively
  Visual Analog Scale (VAS, 0-10; 0= no pain and 10= very severe unbearable pain) at 0-1-2-4-8-12 and 24th hours

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Sertcakacilar, MD, Study Director — Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No